CLINICAL TRIAL: NCT03485417
Title: Substance Misuse To Psychosis for Stimulants (SToP-S)--An Early Assertive Pharmacotherapy Intervention Study
Brief Title: Substance Misuse To Psychosis for Stimulants
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Queen Mary Hospital, Hong Kong (Other); North District Hospital (Other)
Responsible Party: Principal Investigator, Dr. Albert Kar-Kin Chung, Clinical Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SToP-S
Record Dates: First submitted 2018-03-14; First posted 2018-04-02 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Stimulant Use With Stimulant-Induced Psychotic Disorder (Diagnosis); Schizophrenia and Related Disorders; Stimulant Dependence; Stimulant Abuse; Pharmacotherapy
Keywords: stimulant; psychosis; schizophrenia; dependence; pharmacotherapy
MeSH Terms: conditions — Disease; Schizophrenia; Psychotic Disorders | interventions — Aripiprazole; Paliperidone Palmitate; Therapeutics

STUDY DESIGN:
Intervention Model Description: prospective randomised single-blinded
Who Masked: Outcomes Assessor
Masking Description: treatment group randomised to each participant is masked to the outcome assessors
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Aripiprazole Arm (Active Comparator): Aripiprazole (oral or depot) Oral: 10-30mg daily Depot: 300-400mg every four week; Intramuscularly
  Interventions: Drug: Aripiprazole
- Paliperidone Arm (Active Comparator): Paliperidone (oral or depot) Oral: 3-12mg Depot: Intramuscularly; a) sustenna 50-150mg every four weekly, or b) trinza 273-819mg every 12 weekly
  Interventions: Drug: Paliperidone
- Treatment as Usual Arm (Other): Treatment as Usual arm
  Interventions: Other: Treatment as Usual

INTERVENTIONS:
Drug: Aripiprazole — for oral or depot preparation
  Arms: Aripiprazole Arm
Drug: Paliperidone — for oral or depot
  Arms: Paliperidone Arm
Other: Treatment as Usual — to be decided by treating psychiatrist with Rx other than aripiprazole or paliperidone
  Arms: Treatment as Usual Arm

SUMMARY:
In Hong Kong, less than 5% of stimulants abusers were reported to misuse these substances via injection. Also, it is well known that patients with co-morbid substance abuse/dependence and psychosis or schizophrenia-related disorders are prone to earlier treatment discontinuation and high oral medication non-adherence, resulting in poorer overall outcomes. With the recent availabilities of the 4-weekly long-acting injectable form of aripiprazole, and the 4-weekly and the 3-monthly long-acting injectable form of paliperidone palmitate, on the background of the surging phenomenon of stimulant misuses in Hong Kong, it is a timely opportunity to conduct an early pharmacotherapy intervention study to offer an evidence-based strategy aiming to stop individuals with substance use disorders with psychosis to develop into a more chronic disabling dependence or co-morbid state.

ELIGIBILITY:
Inclusion Criteria:

• Stimulant use disorder with psychosis or positive stimulant urine test results twice in a month with psychosis

Exclusion Criteria:

* Age <16 years old
* Unable to read English or Chinese
* Unable to give informed consent
* Had been diagnosed to have Intellectual Disabilities (DSM-5) or Mental Retardation (ICD-10 F70-73)
* Had been diagnosed to have Schizophrenia
* Had been diagnosed to have other substance-induced psychotic or mood disorder, including alcohol
* Had been diagnosed to have bipolar disorder viii. Had been diagnosed to have major depressive disorder with psychotic features
* Had been taking any maintenance dose of oral antipsychotics continuously ≥12 weeks AND with psychotic symptoms in remission
* Had been receiving any maintenance dose of long-acting injectable (LAI/depot) antipsychotics continuously ≥4 month AND with psychotic symptoms in remission
* Had known hypersensitivity to risperidone (oral or LAI), paliperidone (oral or LAI), or aripiprazole (oral or LAI)
* Had known history of tardive dyskinesia
* Had known history of neuroleptic malignant syndrome
* Pregnant
* Mother currently breast-feeding
* Had history of prolonged corrected QT interval (QTc) ≥500ms and/or known unstable or untreated cardiac disorder
* Had mild to severe renal impairment with Glomerular Filtration Rate <80 mililitre /min

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 165 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Efficacy on psychosis as measured by the Brief Psychiatric Rating Scale - 24 items (BPRS-24) | at 12th and at 24th months
  The efficacy for controlling stimulant associated psychosis for subjects receiving the active treatments with paliperidone and aripiprazole as compared to treatment as usual is measured by BPRS. The lowest score of BPRS-24 is 24. The lower the score of BPRS refers to better efficacy in controlling psychosis.

SECONDARY OUTCOMES:
transition from diagnosis of substance induced psychosis to Schizophrenia as defined by DSM-5 | 24 months
  The rate of transition from substance induced psychosis To schizophrenia in all 3 different arms
change in stimulant use disorder as defined by DSM-5 | At 12th month and at 24th month
  The change is severity of the Stimulant Use Disorder in subjects in the 3 different arms by DSM-5 criteria
Montreal Cognitive Assessment (MoCA) | At 12th month and at 24th month
  Difference in cognitive outcome measured using MoCA in subjects randomized to the 3 arms. MoCA has the maximum score of 30. A cut-off score of higher than or equal to 26 refers to normal cognition.
Addiction Severity Index (ASL)-lite | At 12th and 24th months
  Difference in functional outcome measured using ASL-lite in subjects randomized to the 3 treatment arms

CONTACTS AND LOCATIONS:
Overall Officials: albert KK Chung, Dr, Principal Investigator — The University of Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong